CLINICAL TRIAL: NCT02542774
Title: Sex Differences in the Risk of Cardiovascular Diseases Associated With Diabetes: an Examination of Variation in Health Service Delivery
Brief Title: Sex Differences in the Risk of Cardiovascular Diseases Associated With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15_108R
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Stroke; Myocardial infarction; Stable angina pectoris; Heart failure; Quality of care
MeSH Terms: conditions — Diabetes Mellitus; Stroke; Myocardial Infarction; Angina, Stable; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention is given. — This study is based on the analysis of linked electronic health records (CALIBER dataset)

SUMMARY:
To evaluate the risk of cardiovascular events associated with medication use for controlling blood glucose, blood pressure and cholesterol levels in men and women with diabetes treated in primary care

DETAILED DESCRIPTION:
The management and treatment of adult diabetes is far from optimal. The most recent report from the National Diabetes Audit showed that only one in three people with diabetes are achieving recommended standards for controlling blood glucose, blood pressure and cholesterol levels; and only three in five received basic care processes to reduce their risk of diabetes-related complications such as blindness, amputation and kidney disease. Women did 15% worse than men, which may explain some of the reported higher excess risk of coronary heart disease and stroke, consequent to diabetes in women than men. More efficient and equitable care in people with diabetes could lead to substantial cost savings, and would improve the lives of women and men currently living with diabetes.

The objective of this research isto evaluate the risk of cardiovascular events associated with medication use for controlling blood glucose, blood pressure and cholesterol levels in men and women with diabetes treated in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes at or before study entry, and participants who develop new-onset diabetes during follow-up.
* Age ≥ 18 years
* Data collected in the period 1997-2010
* Minimum time since registration of 1 year
* Minimum of 1 year of up to standard data (CPRD quality standard)

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the CALIBER database who have diabetes, are included in the Clinical Practice Research Datalink (CPRD) and consented to data linkage.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
First occurrence of cardiovascular disease | 10 years
  First recorded diagnosis of cardiovascular disease during follow-up: stable angina, unstable angina, myocardial infarction, unheralded coronary death, heart failure, transient ischaemic attack, ischaemic stroke, subarachnoid haemorrhage, intracerebral haemorrhage, peripheral arterial disease, abdominal aortic aneurysm, ventricular arrhythmia, cardiac arrest, or sudden cardiac death

SECONDARY OUTCOMES:
Cardiovascular mortality | 10 years
  Composite endpoint of cardiovascular mortality
All cause mortality | 10 years
  Composite endpoint of all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Peters, Study Director — The George Institute
Locations (1):
- The George Institute for Global Health, Nuffield Department for Population Health, University of Oxford, Oxford, Oxford, United Kingdom